CLINICAL TRIAL: NCT00493974
Title: Antileukotriene Therapy for COPD Exacerbations
Brief Title: Zileuton to Treat Adults With Chronic Obstructive Pulmonary Disease (The LEUKO Study)
Acronym: LEUKO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of feasibility due to low recruitment
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0701M00621; U10HL074424 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Exacerbation; Anti-leukotriene; Length of Stay; LOS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — zileuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zileuton (Active Comparator): Zileuton (Zyflo, 600 mg 4 times a day)
  Interventions: Drug: Zileuton
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zileuton — Zyflo tablets, 600 mg, 4 times a day
  Other Names: Zyflo
  Arms: Zileuton
Drug: Placebo — Placebo 4 x daily
  Other Names: Inactive Matching Placebo
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a long-term lung disease that is caused by cigarette smoking or by breathing in other lung irritants, including pollution, dust, or chemicals. The purpose of this study is to evaluate the effectiveness of zileuton, a medication that is used to control asthma symptoms, at reducing the length of a hospital stay for adults who are hospitalized for a COPD exacerbation, or worsening of COPD symptoms.

DETAILED DESCRIPTION:
COPD is a disease in which the lung airways are partly damaged and obstructed, making it difficult to breathe. COPD is the fourth leading cause of death in the United States. Symptoms include coughing, excess mucus production, shortness of breath, wheezing, and chest tightness. Treatment usually includes inhaled bronchodilator or steroid medications that work by relaxing the muscles around the lung airways and reducing inflammation. Zileuton, a medication that is used to prevent asthma symptoms, may be beneficial in treating people who experience COPD exacerbations. Zileuton works by blocking the formation of substances that cause inflammation, fluid retention, and constriction in the lungs. The purpose of this study is to evaluate the effectiveness of zileuton at reducing the length of a hospital stay for adults who are hospitalized for a COPD exacerbation.

This study will enroll adults who are admitted to the hospital due to severe COPD symptoms. Participants will be randomly assigned to receive either zileuton or placebo four times a day for up to 14 days. While in the hospital, lung function testing and urine collection will occur. Study visits will occur at Days 14 and 30, and will include lung function testing, a medical history review, and a study drug adverse effects review.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital for a COPD exacerbation
* FEV1 less than 60% of predicted level
* At least 10 pack years of smoking

Exclusion Criteria:

* Any uncontrolled systemic disease
* Known hypersensitivity to zileuton
* Asthma
* Lobar pneumonia or pulmonary edema
* Interstitial lung disease
* Medical condition that is likely to limit survival to less than 30 days at the time of study entry
* History of liver disease
* Current use of theophylline
* Participation in another clinical trial in the COPD Clinical Research Network
* Incarceration
* Institutionalization
* Pregnant
* History of a suicide attempt
* Prior inpatient admission for a psychiatric disorder
* Bipolar disorder

'

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prescott Woodruff, MD, Study Chair — University of California at San Francisco
Locations (18):
- United States (18):
  - University of Alabama Lung Health Center, Birmingham, Alabama
  - Veteran's Administration Medical Center, Birmingham, Alabama
  - LA BioMed at Harbor, University of California, Los Angeles, California
  - University of California San Francisco-Airway Clinical Research Center, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - Veteran's Administration Medical Center, Denver, Colorado
  - University of Maryland Hospital, Baltimore, Maryland
  - Fallon Clinic, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Veteran's Administration Medical Center, Boston, Massachusetts
  - Veteran's Administration Medical Center, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Veteran's Administration Medical Center, Minneapolis, Minnesota
  - HealthPartners Research Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Emphysema Research Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodruff PG, Albert RK, Bailey WC, Casaburi R, Connett JE, Cooper JA Jr, Criner GJ, Curtis JL, Dransfield MT, Han MK, Harnden SM, Kim V, Marchetti N, Martinez FJ, McEvoy CE, Niewoehner DE, Reilly JJ, Rice K, Scanlon PD, Scharf SM, Sciurba FC, Washko GR, Lazarus SC; Copd Clinical Research Network. Randomized trial of zileuton for treatment of COPD exacerbations requiring hospitalization. COPD. 2011 Feb;8(1):21-9. doi: 10.3109/15412555.2010.540273. PMID 21299475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ER's and inpatient units from 10 main clinical sites (and their affiliated hospitals) between September 2007 and October 2008.
Pre-assignment Details: Participants were screened using the eligibility criteria before randomization.
Groups:
- Placebo: Matching placebo 4 times a day
Period: Overall Study
Arm/Group | Zileuton | Placebo
Started | 60 | 59
Completed | 47 | 45
Not Completed | 13 | 14
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zileuton | Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.2) | 64.3 (9.5) | 63.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 56 | 57 | 113
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All applicable categories were checked for each participant.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 16 | 24 | 40
    White | 36 | 31 | 67
    More than one race | 7 | 3 | 10
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Admission will begin at the time the subject has been admitted to an inpatient service. Length of Stay (LOS) will be recorded in days. The LOS will be based on the number of days spent in an acute medical ward or in the ICU. Subjects that are admitted and discharged in the same 24 hour period will be recorded as a LOS of 1 day, as will subjects discharged in the ensuing 24 hour period. LOS's greater than 10 days will be truncated to 10 days.
Time Frame: Measured at Day 30
Population: Participants were analyzed following intention to treat (ITT) method.
  One participant randomized to Zileuton withdrew consent before hospital discharge.
  Days to discharge are set at a maximum of 10 days.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 59 | 59
Days | 3 (2.19) | 3 (3.06)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = .3876, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in FEV1% Predicted
Description: Change in Post-bronchodilator FEV1% predicted comparing data at 30 day visit with baseline.
Time Frame: Measured at Baseline and Day 30
Population: Participants were analyzed using the intent to treat method. The N is lower than total randomized due to participants that were unable to perform spirometry at baseline.
Measure: Mean (Standard Error); unit: percent predicted
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 14 | 9
percent predicted | 6.8 (4.2) | 8.0 (4.4)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = 0.6413, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in FEV1/FEV6 Levels
Description: Change in Post-bronchodilator FEV1/FEV6 ratio comparing data at discharge visit with baseline.
Time Frame: from baseline to day of discharge
Population: Participants were analyzed using the intent to treat method. The N is lower than total randomized due to participants that were unable to perform spirometry at baseline and missing discharge data.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 8 | 8
ratio | 0.02 (0.03) | 0.03 (0.02)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = 0.6433, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Treatment Failure
Description: Treatment failure is defined as death, intubation, readmission to a hospital for COPD, urgent visit to an outpatient or ED provider for symptoms of COPD or intensification of therapy [including second course of antibiotics for COPD, and second course of systemic steroids for COPD]) in the first 30 days after randomization.
Time Frame: Baseline to day 30 visit
Population: Participants were analyzed following intention to treat (ITT) method.
Measure: Number; unit: Participants
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 60 | 59
Participants
  Death | 1 | 2
  Intubation | 1 | 1
  Hospital Readmission | 7 | 7
  Urgent Visit | 7 | 6
  Intensification of therapy | 11 | 11
  Any Treatment Failure | 14 | 16
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = 0.63, Chi-squared

5. Secondary Outcome: Health-related Quality of Life
Description: St. George's Respiratory Questionnaire - Total Score
  The SGRQ was asked with respect to the last one month as validated for acute exacerbations of COPD by Doll et al.
  Scale from 0 (no disability) to 100 (maximum disability).
  The SGRQ total score summarizes the impact of airway specific disease on overall health status. Scores range from zero (no impairment) to 100 (maximum impairment). Scores were calculated using the SGRQ scoring Algorithm.
Time Frame: Change from Baseline and 1 Month
Population: Participants were analyzed using the intent to treat method and included those that had SGRQ data at baseline and 1 month.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 46 | 43
Units on a scale | -10.6 (14.8) | -8.5 (14.6)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = 0.4957, t-test, 2 sided

6. Secondary Outcome: Change in Urinary Leukotriene (LTE4) Levels
Description: Change in natural log-transformed LTE4 (ng/mg Cr.) from Baseline to 24 Hours
Time Frame: Baseline and 24 hours
Population: Intent to Treat.
  Participants with urine sample at both visits.
Measure: Log Mean (Standard Error); unit: (ng/mg Cr.)
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 46 | 42
(ng/mg Cr.) | -1.38 (0.17) | 0.14 (0.22)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: Change in Urinary Leukotriene (LTE4) Levels
Description: Change in natural log-transformed LTE4 (ng/mg Cr.) from Baseline to 72 Hours
Time Frame: Baseline and 72 hours later
Population: Intent to Treat.
  Participants with urine sample at both visits.
Measure: Log Mean (Standard Error); unit: (ng/mg Cr.)
Arm/Group | Zileuton | Placebo
Number analyzed (Participants) | 22 | 20
(ng/mg Cr.) | -1.32 (0.40) | 0.26 (0.38)
Statistical Analysis 1: Comparison: Zileuton vs Placebo; Test type: Superiority or Other; p = 0.006, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events from randomization to the 30 day follow-up visit. AEs that continued past the end of the study period were followed until the Investigator believed it reached a stable clinical endpoint or resolved.
Arm/Group | Zileuton | Placebo
Serious Adverse Events (participants affected / at risk) | 17/60 | 20/59
Other Adverse Events (participants affected / at risk) | 13/60 | 12/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zileuton (N=60) | Placebo (N=59)
Allergic Reaction( to amiodarone) (Immune system disorders) | 1 (1) | 0 (0)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Depressive disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MRSA bursitis (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium Avium Intracellular Complex (Infections and infestations) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zileuton (N=60) | Placebo (N=59)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19) | 6 (14)
COPD worsening (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects recruited

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No